CLINICAL TRIAL: NCT00407199
Title: The Use of Quetiapine (Seroquel) in the Treatment of Social Phobia: Effects on Cue Reactivity in Response to Virtual Reality Public Speaking Environment
Brief Title: The Use of Quetiapine (Seroquel) in the Treatment of Social Phobia: Public Speaking Environment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0608M91257; M91527
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Social Phobia
Keywords: social phobia, anxiety, quetiapine
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: quetiapine

SUMMARY:
This is a pilot study that will focus on the collection of preliminary data to determine the efficacy of quetiapine for individuals with social phobia. We hypothesize that individuals will react with less self-reported anxiety and physiological reactivity in the drug condition than in the placebo condition. If true, this would constitute a strong signal for a significant treatment effect for quetiapine in social phobia. A positive treatment effect in this study would provide rationale for further investigation of the efficacy of quetiapine for cue reactivity for individuals with social phobia. Further study would include increased sample size in order to obtain statistical power and replication of findings. We will utilize the IR formulation of quetiapine.

DETAILED DESCRIPTION:
Primary Objective:

The purpose of this study is to evaluate the use of quetiapine to diminish cue reactivity to a Virtual Reality environment for individuals with Social Phobia. The following primary and secondary outcome measures will be administered to subjects during each Virtual Reality exposure in treatment and non-treatment conditions. The outcome measures have demonstrated adequate reliability and validity in the detection of clinical change for individuals with social phobia in open label studies using quetiapine (Schutters, van Megen, and Westenberg, 2005). The Personal Report of Confidence as a Speaker (PRCS; Paul, 1966) will be utilized as the primary measure to establish individual diagnosis and severity level. Pertaub and Slater (2002) demonstrated the sensitivity of the PRCS in measuring anxiety responses to virtual audiences. A total score of 21 or greater on the PRCS will be required for study inclusion (Carrigan and Levis, 1999). Carrigan and Lewis (1999) reported a mean score of 23.73 on the 30-item PRCS for individuals reporting fear of public speaking. Subjective units of distress ratings and measures of blood pressure and heart rate will be obtained within session in order to measure immediate changes in subject's cue reactivity to VRE stimuli. The outcome measures include:

Primary Measure: Personal Report of Confidence as a Speaker (PRCS)

Secondary Measures:

Liebowitz Social Anxiety Scale (LSAS) Clinical Global Impressions-Improvement Scale (CGI) Brief Social Phobia Scale Social Phobia Inventory Fear of Negative Evaluation Scale Hamilton Rating Scale for Anxiety In session-Subjective Units of Distress Blood Pressure and heart rate monitored within session

Design:

A crossover, double-blind within subjects design will be used. The two conditions are placebo and drug prior to exposure to social anxiety cues in the virtual environment. Each subject will be in both conditions over the course of two visits. Each subject will be in only one condition on the first visit and will then cross-over to the other condition on the second visit. Order will be counter-balanced across subjects. The treatment phase of the study will include the two afore mentioned visits, totaling 60 minutes each. This will include the treatment and pre-post assessment

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* Primary DSM-IV Axis I diagnosis of social phobia, specific fear of public speaking
* PRCS total score: 21 or greater (1 SD above population norm of 14.2)

Exclusion Criteria:

* Current contraindications/sensitivity to quetiapine
* Current prescription of benzodiazepine, tranquilizer, or antipsychotic medication
* Current Psychotic episode
* Current Manic episode
* Current Depressive episode
* Current drug or alcohol dependence
* A patient with diabetes mellitus (DM) fulfilling one of the following criteria:

  * Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) 8.5%.
  * Admitted to hospital for treatment of DM or DM related illness within the past 12 weeks
  * Not under physician care for DM.
  * Physician responsible for patient's DM care has not indicated that the patient's DM is controlled.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Personal Report of Confidence as a Speaker (PRCS)

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS)
Brief Social Phobia Scale
Social Phobia Inventory
Fear of Negative Evaluation Scale
In session-Subjective Units of Distress
Blood Pressure and heart rate monitored within session

CONTACTS AND LOCATIONS:
Overall Officials: David E Adson, M.D., Principal Investigator — University of Minnesota; Christopher B Donahue, Ph.D., Principal Investigator — Univeristy of Minnesota; Matt Kushner, Ph.D. LP, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Donahue CB, Kushner MG, Thuras PD, Murphy TG, Van Demark JB, Adson DE. Effect of quetiapine vs. placebo on response to two virtual public speaking exposures in individuals with social phobia. J Anxiety Disord. 2009 Apr;23(3):362-8. doi: 10.1016/j.janxdis.2008.12.004. Epub 2008 Dec 24. PMID 19157776